CLINICAL TRIAL: NCT04071106
Title: Turmeric Based Therapy in the Treatment of Psoriasis: A Clinical Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hagar Nofal, Assistant Lecturer, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#3950-20-8-2017
Record Dates: First submitted 2019-08-14; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Turmeric; Curcumin; Olive oil; Dermoscopy; NFkB
MeSH Terms: conditions — Psoriasis | interventions — turmeric extract; Olive Oil; Petrolatum; calcipotriene; Betamethasone

STUDY DESIGN:
Intervention Model Description: Five groups will be included in the study Group 1: 10 Psoriatic patients receive turmeric extract based ointment . Group 2: 10 psoriatic patients will receive turmeric extract + olive oil based ointment.
  Group 3: 10 psoriatic patients will receive petrolatum base as negative control.
  Group 4: 10 psoriatic patients will receive NBUVB as positive control. Group 5: 10 psoriatic patients will receive established topical treatment serving as 2nd positive control.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients do not know whether they are receiving the drugs with active ingredients or negative control. The pathologist will be masked regarding the groups and the point of time before or after therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Turmeric Extract group (Active Comparator): 10 psoriasis patients receiving turmeric based ointment levigated in glycerin twice daily and assessed for response and side effects weekly for 12 weeks
  Interventions: Drug: Turmeric Extract
- Turmeric extract + olive oil group (Active Comparator): 10 psoriasis patients receiving turmeric extract levigated in olive oil instead of glycerin. The ointment will be applied twice daily for 12 weeks & will be assessed weekly
  Interventions: Drug: Turmeric Extract in Olive oil
- Petrolatum group (Placebo Comparator): 10 Psoriasis patients will receive the base of the therapeutic ointment which is the petrolatum. Patients will apply it twice daily and will be assessed weekly clinically and dermoscopically for 12 weeks
  Interventions: Drug: Petrolatum
- NBUVB group (Active Comparator): 10 Psoriasis patients will receive two sessions of NBUVB weekly for 12 weeks and will be assessed weekly clinically and with dermoscope.
  Interventions: Device: NB-UVB
- Established ttt group (Active Comparator): 10 Psoriasis patients will receive topical betamethasone dipropionate or calcipotriol cream twice daily for 12 weeks and will be assessed on weekly basis clinically and by dermoscope
  Interventions: Drug: calcipotriol/ Betamethasone

INTERVENTIONS:
Drug: Turmeric Extract — Patient will apply the treatment twice daily for 12 weeks and will be assessed clinically and by dermoscope weekly and by histopathology every 4 weeks
  Arms: Turmeric Extract group
Drug: Turmeric Extract in Olive oil — Patient will apply the treatment twice daily for 12 weeks and will be assessed clinically and by dermoscope weekly and by histopathology every 4 weeks
  Arms: Turmeric extract + olive oil group
Drug: Petrolatum — Patient will apply the treatment twice daily for 12 weeks and will be assessed clinically and by dermoscope weekly and by histopathology every 4 weeks
  Arms: Petrolatum group
Device: NB-UVB — Patients will receive 2 sessions of NB-UVB phototherapy and will be assessed clinically and by dermoscope weekly and by histopathology every 4 weeks
  Arms: NBUVB group
Drug: calcipotriol/ Betamethasone — Patient will apply the treatment twice daily for 12 weeks and will be assessed clinically and by dermoscope weekly and by histopathology every 4 weeks
  Arms: Established ttt group

SUMMARY:
Psoriasis affects around 4% of world population. The disease could be disabling and disfiguring dermatologic condition. World Health Organization (WHO) has recently drawn the attention to the inadequate treatment options psoriasis patients suffer from among other problems. Furthermore, the available treatment options have many side effects. A lot of the effective treatment options are either expensive or not appropriate for hepatic patients who represent a large subset of Egyptian psoriatic patients. This highlights the need for inexpensive and safe alternative. The effectiveness of Turmeric in psoriasis treatment have been addressed in few reports. Having an immune modulatory effect especially as anti NFκB it is expected to be effective therapy with minimal side effect. Up to the investigator's knowledge this is the first study addressing the efficacy of combined turmeric and olive oil based topical therapy in psoriasis treatment

DETAILED DESCRIPTION:
Psoriasis is a prevalent skin disorder. It affects around 4% of world's population. It can be disfiguring and disabling in severe cases. There is dysregulated immune response in psoriatic patients to unknown injurious agents with upregulation of Th1/Th17 pathways which is mediated via Nuclear Factor kappa B (NFκB). NFκB is a key player in psoriasis development; its activation and nuclear translocation is present in every step of the way of psoriasis starting from keratinocyte release of cytokines -in response to stress- to the maturation and activation of dendritic cells, to the continuous loop of T cell activation.

Turmeric extract has anti-inflammatory, anti-oxidant, anti-microbial and anti-carcinogenic effects. It has inhibitory effects on NF-κB and various cytokines production.

In this clinical trial 5 groups of patients with mild to moderate psoriasis are recruited; group (A) Receiving the Turmeric extract based ointment only. Group (B) receiving Turmeric extract + olive oil based treatment. Group (C) will serve as negative control receiving only petrolatum base. Group (D) will receive NB UVB serving as positive control. Group (E) will receive established topical treatment serving as positive control.

Each patient will be assessed on weekly bases clinically for the disease severity using PASI score and via dermatoscope. Histopathological evaluation (H& E along with NFkB expression analysis) will be done at 4 points of time baseline, 4 weeks, 8 weeks, 12 weeks through the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mild to moderate psoriasis vulgaris of any age & gender.
2. Patient didn't receive any systemic or topical therapy for psoriasis the last 4 weeks.

Exclusion Criteria:

1. Patients previously received topical or systemic therapy for psoriasis in the past 4 weeks.
2. Patients with pustular or erythrodermic psoriasis.
3. Patients with other dermatological diseases.
4. Patients have hypersensitivity from the active ingredients of the therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area & Severity Index (PASI) | 12 weeks
  Response to therapy is assessed via measurement of (PASI) every week for 12 w. The range of PASI score is from 0 (no disease) - 72 (sever disease). In PASI, the body is divided into four sections (head; arms; trunk; legs). Each of the sections is scored by itself, and then the four scores are combined into the final PASI. For each section, area of involved skin is given a grade from 0 to 6: 0= 0% of involved area, 1 = < 10% involved, 2=10-29% involved, 3 =30-49% involved area, 4 = 50-69% involved, 5 =70-89% involved, 6 = 90-100%involved. Within each section, the severity is estimated in three clinical parameters: erythema (redness), induration (thickness) and desquamation (scaling). Severity parameters are measured on a scale of 0 to 4, from none to maximum. The sum of three severity parameters is calculated for each section of body, multiplied by the area score for that section and multiplied by weight of respective section (0.1 for head, 0.2 for arms, 0.3 for body and 0.4 for legs).
Change on pathology level | Baseline and every 4 weeks for the period of the study (12 w)
  Histopathologic evaluation of hematoxylin and eosin stained slides from psoriatic lesions before and after treatment or placebo. The slides will be given a score based on the presence or absence of each of the following: Hyperkeratosis (0.5), One mitosis/3 rete ridges (0·5), Acanthosis (1),Dermis lymphocytic infiltrate; Mild (0·5) Moderate (1) Marked (2·0) Parakeratosis (1),Papillary congestion (0.5),Lack of granular layer (1), Munro abscesses (2), Thinning above the papillae (0.5), Length of rete ridges (0.5), Clubbing of rete ridges (0·5). The sum score of each patient's slide will be recorded at baseline & every 4 week
Change in NFϰB expression | Baseline and every 4 weeks till the end of 12 weeks.
  The NFϰB expression will be identified by the percentage of positive nuclear stained epidermal cells in slide at base line and every 4 weeks till the end of study which is 12 week
Change in psoriasis severity | Weekly basis for 12 weeks
  Response to therapy will be assessed using dermatoscope with software mediated image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Nofal, Principal Investigator — Assistant lecturer

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, Analytic Code
Time Frame: 2 Years after the finish of the study

REFERENCES:
- [Background] Avramidis G, Kruger-Krasagakis S, Krasagakis K, Fragiadaki I, Kokolakis G, Tosca A. The role of endothelial cell apoptosis in the effect of etanercept in psoriasis. Br J Dermatol. 2010 Nov;163(5):928-34. doi: 10.1111/j.1365-2133.2010.09935.x. PMID 20633014
- [Background] Cai Y, Fleming C, Yan J. Dermal gammadelta T cells--a new player in the pathogenesis of psoriasis. Int Immunopharmacol. 2013 Jul;16(3):388-91. doi: 10.1016/j.intimp.2013.02.018. Epub 2013 Mar 13. PMID 23499509
- [Background] Camacho-Barquero L, Villegas I, Sanchez-Calvo JM, Talero E, Sanchez-Fidalgo S, Motilva V, Alarcon de la Lastra C. Curcumin, a Curcuma longa constituent, acts on MAPK p38 pathway modulating COX-2 and iNOS expression in chronic experimental colitis. Int Immunopharmacol. 2007 Mar;7(3):333-42. doi: 10.1016/j.intimp.2006.11.006. Epub 2006 Dec 18. PMID 17276891
- [Background] Coimbra S, Figueiredo A, Castro E, Rocha-Pereira P, Santos-Silva A. The roles of cells and cytokines in the pathogenesis of psoriasis. Int J Dermatol. 2012 Apr;51(4):389-95; quiz 395-8. doi: 10.1111/j.1365-4632.2011.05154.x. PMID 22435425
- [Background] Goldminz AM, Au SC, Kim N, Gottlieb AB, Lizzul PF. NF-kappaB: an essential transcription factor in psoriasis. J Dermatol Sci. 2013 Feb;69(2):89-94. doi: 10.1016/j.jdermsci.2012.11.002. Epub 2012 Nov 14. PMID 23219896

DOCUMENTS (1):
  • Study Protocol (2019-08-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT04071106/Prot_000.pdf